CLINICAL TRIAL: NCT01592110
Title: A Pilot, Open-Label, Non-Randomized, Single Ascending Dose, Safety and Pharmacokinetic Trial With Injectable Risperidone-SABER and the DosePro Delivery System in Patients With Chronic, Stable Schizophrenia or Schizoaffective Disorder
Brief Title: A Safety and PK Study of Injectable Risperidone-SABER and the DosePro Delivery System in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZX003-1101
Record Dates: First submitted 2012-05-01; First posted 2012-05-07 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 25 mg of risperidone-SABER administered as a SC injection of 0.25 mL (100 mg/mL concentration) in the abdominal region
  Interventions: Drug: risperidone-SABER
- Cohort 2 (Experimental): 50 mg of ZX003 (risperidone-SABER-DosePro) administered as 0.5 mL (100 mg/mL concentration) via the DosePro Needle-free Delivery System in the abdominal region
  Interventions: Other: ZX003:risperidone-SABER and the DosePro System
- Cohort 3 (Experimental): 50 mg of risperidone-SABER administered as a SC injection of 0.5 mL (100 mg/mL concentration) in the abdominal region
  Interventions: Drug: risperidone-SABER
- Cohort 4 (Experimental): 100 mg of risperidone-SABER administered as a SC injection of 1.0 mL (100 mg/mL concentration) in the abdominal region
  Interventions: Drug: Risperidone-SABER

INTERVENTIONS:
Drug: risperidone-SABER — 25 mg of risperidone-SABER administered as a subcutaneous (SC) injection of 0.25 mL
  Arms: Cohort 1
Other: ZX003:risperidone-SABER and the DosePro System — 50 mg risperidone-SABER administered as 0.5 mL via the DosePro Needle-Free Injection System
  Arms: Cohort 2
Drug: risperidone-SABER — 50 mg of risperidone-SABER administered as a SC injection of 0.5 mL
  Arms: Cohort 3
Drug: Risperidone-SABER — 100 mg of risperidone-SABER administered as a SC injection of 1.0 mL
  Arms: Cohort 4

SUMMARY:
This is a Phase 1, open-label study to evaluate the safety and pharmacokinetics (PK) of three doses of risperidone-SABER, administered with a needle and syringe or via the DosePro Needle-Free Delivery System in patients with chronic, stable schizophrenia.

DETAILED DESCRIPTION:
This is an open-label, single ascending dose (SAD), safety and PK study in patients with chronic, stable schizophrenia or schizoaffective disorder. Patients will participate in the study for a total of up to 10 weeks for Cohorts 1-3, including a Screening period of up to 35 days and a study treatment period of 35 days, and up to 14 weeks for Cohort 4, including a Screening period of up to 35 days and a study treatment period of 63 days. Patients will be assigned to one of four cohorts, and will receive a single dose of 25 mg, 50 mg or 100 mg (100 mg/mL concentration) administered as a single subcutaneous (SC) injection or via the DosePro Needle-Free Delivery System.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older.
* Diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder as per DSM-IV criteria in the past 6 months or more, dependent on diagnosis.
* Currently on maintenance antipsychotic medication (i.e., patients treated with antipsychotic medication with stable doses in the 4 weeks prior to Screening and no psychosis-related dose changes in the 8 weeks prior to Screening).
* Body Mass Index (BMI) (kg/m2) ≥ 20 and ≤ 40.
* Female patients with:

  * Non-childbearing potential (surgically sterile [hysterectomy]) or post-menopausal ≥ 2 years -OR-
  * Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (hormonal contraception, abstinence, diaphragm with spermicide, condom with spermicide, or intrauterine device) from Screening until the End-of-Study visit.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in the 12-lead electrocardiogram (ECG).
* No clinically significant findings from a vital signs measurement.
* Be informed of the nature of the study and give written consent prior to initiating any study procedure.

Exclusion Criteria:

* Have known or suspected carcinoma.
* Have known presence or history of renal or hepatic insufficiency.
* Have known history, hypersensitivity or idiosyncratic reaction (including dystonias) to risperidone, paliperidone, and/or any other drug substance with similar activity.
* Have a history of alcohol or drug-dependence as per DSM-IV criteria during the 6-month period immediately prior to Screening.
* Have a history of epilepsy or risk of having seizures.
* Are pregnant, lactating, or likely to become pregnant during the study.
* Have taken an antipsychotic depot product (including investigational products) within the 60 days prior to Screening.
* Participated in another clinical trial or received an investigational product within 30 days prior to Screening.
* Have a positive alcohol breathalyzer test at Screening or Admission.
* Have a positive Screening test for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Have a positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, etc.) at Screening or Admission.
* Excessive use of caffeine-containing beverages exceeding 500 mg caffeine/day (5 cups of coffee).
* Are unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to Admission until End-of-Study.
* Excessive smoking as judged by the Investigator
* Donation of blood (> 500 mL) or blood products within 2 months (56 days) prior to Admission.
* Have used any concomitant medications significantly impacting CYP2D6 (moderate and strong inducers/inhibitors), including but not limited to those outlined in Appendix 1, within 14 days or 5 half-lives (whichever is longer) prior to Admission. Medications judged to not interact with risperidone may be continued at the discretion of the Investigator and in accordance with the protocol requirements for tapering and wash-out.
* Are unwilling to abstain from vigorous exercise (as judged by the Investigator) from 48 hours prior to Admission until End-of-Study.
* Are unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study.
* Are unlikely to comply with the protocol requirements, instructions and study- related restrictions (e.g., uncooperative attitude, inability to return for out-patient visits or improbability of completing the clinical study).
* Have previously been enrolled in this clinical study.
* Are unable to tolerate the oral risperidone challenge on Screening Day -3.
* Are unable to stabilize on antipsychotic medication tapering during the Screening period.

Note that "Admission" in the above criteria refers to Admission and Qualification which occurs on day -4 for Cohort 1 and Day -6 for Cohorts 2 and 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number and percent of patients experiencing a treatment emergent adverse event following a single dose of risperidone-SABER | Within 35 days post-dose
Maximum plasma concentration, time of maximum plasma concentration and area under the concentration time curve for risperidone, 9-OH risperidone and active moiety (risperidone + 9-OH risperidone) | Within 35 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Lev G Gertsik, MD, Principal Investigator — Parexel
Locations (1):
- Glendale Adventist Medical Center, Glendale, California, United States